CLINICAL TRIAL: NCT02769208
Title: Influence of Indoor Air Filtration Strategies on Occupant Health Indicators
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Feng Li (Other)
Collaborators: Duke University (Other); Tsinghua University (Other); Rutgers University (Other)
Responsible Party: Sponsor-Investigator, Feng Li, Attending Physician, Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine
Organization: Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2014KY107
Record Dates: First submitted 2016-05-10; First posted 2016-05-11 (Estimated); Last update posted 2016-06-01 (Estimated); Status verified 2016-05

CONDITIONS: Risk Factors for Respiratory and Cardiovascular Disease
Keywords: Air Pollution; Air Filtration; Exposure Assessment; HEPA Filter; Electrostatic Precipitator; Cardiovascular Disease Biomarkers; Respiratory Disease Biomarkers
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group A: Pre-Filter Only Intervention (Active Comparator): Subjects in Group A start with baseline conditions of pre-filter + HEPA + ESP in their offices and dorms. After a baseline biological measurement, they then receive a 5-week intervention in which both the HEPA and ESP are removed, leaving only a pre-filter. This intervention period includes a biological measurement 2 weeks into the intervention and other 4-5 weeks into the intervention. The baseline air purification conditions are then restored, and another biological measurement is taken 2 weeks after that.
  Interventions: Device: Central air handling unit air purification technologies
- Group B: Pre-filter + HEPA Intervention (Active Comparator): Subjects in Group B start with baseline conditions of pre-filter + HEPA + ESP in their offices and dorms. After a baseline biological measurement, they then receive a 5-week intervention in which the ESP is removed, leaving a pre-filter + HEPA combination. This intervention period includes a biological measurement 2 weeks into the intervention and other 4-5 weeks into the intervention. The baseline air purification conditions are then restored, and another biological measurement is taken 2 weeks after that.
  Interventions: Device: Central air handling unit air purification technologies

INTERVENTIONS:
Device: Central air handling unit air purification technologies — As described in the arm descriptions, the interventions involve changing the baseline pre-filter + HEPA + ESP conditions by removing either just the ESP or both the ESP and the HEPA for a five week period.
  Other Names: Pre-filter; HEPA filter; Electrostatic precipitator (ESP)

SUMMARY:
The purpose of this study is to evaluate whether two different central air purification technologies reduce air pollutant exposure and beneficially influence health as evaluated with a suite of biological markers related to cardiovascular and respiratory disease risk.

DETAILED DESCRIPTION:
This study will test two common types of central air handling unit filtration technologies, high-efficiency particulate air (HEPA) filters and electrostatic precipitators (ESPs), to evaluate the impacts of these technologies on personal exposure to air pollutants and the associated cardiovascular and respiratory health outcomes. HEPA filters remove a high percentage of the particulate matter in the air, as do ESPs, but ESPs also generate ozone, which may have its own detrimental health effects. These air purification technologies will be placed in different combinations with a coarse pre-filter to protect the air exchange machinery (combinations: pre-filter only, pre-filter + HEPA, and pre-filter + HEPA + ESP) in both the residences and offices of study participants living on a factory campus in Changsha, Hunan Province, China. Large dormitories and office buildings with central air handling units are common in China and around the world, and so adding air purification into the central ducts represents a practical strategy to reducing personal exposure to air pollution and related health outcomes. The Changsha area commonly suffers from high air pollution, and the dormitories and offices on this workspace are already outfitted with both HEPA filters and ESPs. Therefore, testing these technologies in this environment presents a natural experimental condition to test the benefits of air purification. The study investigators hypothesize that both the pre-filter + HEPA and pre-filter + HEPA + ESP conditions will reduce particulate matter exposure and reduce biological markers of cardiovascular and respiratory disease compared to the pre-filter alone, but that the ESP will generate enough ozone to lead to lower health benefits than HEPA+pre-filter condition.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults;
* Live and work at the Broad Town work campus in eastern Changsha, Hunan Province, China

Exclusion Criteria:

* Has any of the following diseases: chronic respiratory, cardiovascular, liver, renal, hematological disease; diabetes mellitus;
* Has any other diseases that may confound or complicate the effects of the intervention
* Pregnant females

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 89 (Actual)
Dates: Start 2014-11; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Change from baseline FEV1 | At baseline, 2 weeks and 4 weeks into the intervention period, and then 2 weeks post-intervention
  FEV1 (forced expiratory volume in the first second of exhalation, unit: liter) was measured by spirometry in all subjects at four separate time points to compare FEV1 changes at different times before, during, and after the filtration intervention as a marker of lung function.
Change from baseline soluble P-selectin | At baseline, 2 weeks and 4 weeks into the intervention period, and then 2 weeks post-intervention
  Soluble P-selectin (a protein shed by activated platelets in the blood, unit: ng/ml) was measured by ELISA in plasma in all subjects at four separate time points to compare levels at different times before, during, and after the filtration intervention as a marker of platelet activation.
Change from baseline von Willebrand factor (VWF) | At baseline, 2 weeks and 4 weeks into the intervention period, and then 2 weeks post-intervention
  VWF (a glycoprotein released by damaged vascular cells into the blood, unit: ug/ml) was measured by ELISA in plasma in all subjects at four separate time points to compare levels at different times before, during, and after the filtration intervention as a marker of endothelial cell damage.
Change from baseline augmentation index (AI) | At baseline, 2 weeks and 4 weeks into the intervention period, and then 2 weeks post-intervention
  AI (a measure of how much the reflecting pulse wave augments the outgoing systole pulse wave, unit: N/A (index)) was measured by pulse wave analysis in all subjects at four separate time points to compare levels at different times before, during, and after the filtration intervention as a marker of arterial stiffness.
Change from baseline systolic blood pressure (SBP) | At baseline, 2 weeks and 4 weeks into the intervention period, and then 2 weeks post-intervention
  Brachial SBP (unit: mm Hg) was measured by an oscillometric method in all subjects at four separate time points to compare levels at different times before, during, and after the filtration intervention as a marker of vasoconstriction.
Change from baseline fractional exhaled nitric oxide (FeNO) | At baseline, 2 weeks and 4 weeks into the intervention period, and then 2 weeks post-intervention
  FeNO (produced from inflammatory nitric oxide signalling in the lung, unit: ppb) was measured with an ambient NO-scrubbing collection method and chemiluminescence in all subjects at four separate time points to compare levels at different times before, during, and after the filtration intervention as a marker of airway inflammation.

SECONDARY OUTCOMES:
Change from baseline C-reactive protein (CRP) | At baseline, 2 weeks and 4 weeks into the intervention period, and then 2 weeks post-intervention
  CRP (an inflammatory protein in the blood, unit: ng/ml) was measured with an ELISA in blood samples for all subjects at four separate time points to compare levels at different times before, during, and after the filtration intervention as a marker of systemic inflammation.
Change from baseline 8-hydroxy-2'-deoxyguanosine (8-OHdG) | At baseline, 2 weeks and 4 weeks into the intervention period, and then 2 weeks post-intervention
  8-OHdG (a product of DNA oxidation found in the urine, unit: ng/ml) was measured with LC-MS in urine samples for all subjects at four separate time points to compare levels at different times before, during, and after the filtration intervention as a marker of systemic oxidative stress.
Change from baseline exhaled breath condensate malondialdehyde (EBC MDA) | At baseline, 2 weeks and 4 weeks into the intervention period, and then 2 weeks post-intervention
  EBC MDA (a product of lipid oxidation found in the exhaled breath, unit: nM) was measured with HPLC in exhaled breath condensate samples for all subjects at four separate time points to compare levels at different times before, during, and after the filtration intervention as a marker of airway oxidative stress.
Change from baseline exhaled breath condensate nitrite + nitrate (EBCNN) | At baseline, 2 weeks and 4 weeks into the intervention period, and then 2 weeks post-intervention
  EBCNN (a product of airway inflammatory NO signaling found in the exhaled breath, unit: uM) was measured with HPLC in exhaled breath condensate samples for all subjects at four separate time points to compare levels at different times before, during, and after the filtration intervention as a marker of airway inflammation.
Change from baseline exhaled breath condensate pH (EBC pH) | At baseline, 2 weeks and 4 weeks into the intervention period, and then 2 weeks post-intervention
  EBC pH (a characteristic of exhaled breath associated with inflammation, unit: pH) was measured with a pH meter in exhaled breath condensate samples for all subjects at four separate time points to compare levels at different times before, during, and after the filtration intervention as a marker of airway inflammation.
Change from baseline diastolic blood pressure (DBP) | At baseline, 2 weeks and 4 weeks into the intervention period, and then 2 weeks post-intervention
  DBP (unit: mm Hg) was measured with an oscillometric method for all subjects at four separate time points to compare levels at different times before, during, and after the filtration intervention as a marker of vasoconstriction.
Change from baseline forced vital capacity (FVC) | At baseline, 2 weeks and 4 weeks into the intervention period, and then 2 weeks post-intervention
  FVC (unit: liter) was measured with spirometry for all subjects at four separate time points to compare levels at different times before, during, and after the filtration intervention as a marker of airway function.

CONTACTS AND LOCATIONS:
Overall Officials: Junfeng Zhang, PhD, Principal Investigator — Duke University; Yinping Zhang, PhD, Principal Investigator — Tsinghua University
Locations (1):
- Shanghai First People's Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No